CLINICAL TRIAL: NCT02324764
Title: Use of Glidesheath Slender to Reduce Radial Artery Occlusion and Vascular Access Site Complications Following Transradial Coronary Angiography
Acronym: CAPITAL-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Aun Yeong Chong, Interventional Cardiologist, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20140262
Record Dates: First submitted 2014-12-08; First posted 2014-12-24 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Embolism and Thrombosis of the Radial Artery; Coronary Heart Disease
Keywords: transradial coronary angiography; radial artery occlusion; coronary heart disease; Glidesheath Slender
MeSH Terms: conditions — Embolism; Coronary Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glidesheath Slender (Experimental): The transradial procedure will be performed using the glidesheath slender (studied sheath)
  Interventions: Device: Glidesheath Slender
- Standard sheath (Active Comparator): The transradial procedure will be performed using the standard 6- French radial sheath (comparator sheath)
  Interventions: Device: standard 6- French radial sheath

INTERVENTIONS:
Device: Glidesheath Slender — testing the efficacy and safety of the new transradial sheath in comparison to the standard 6 french sheath.
  Other Names: Glidesheath Slender, Terumo, Tokyo, Japan
  Arms: Glidesheath Slender
Device: standard 6- French radial sheath
  Arms: Standard sheath

SUMMARY:
The objective of this study is to determine the rate of radial artery occlusion and vascular access site complications following transradial angiogram using a new Terumo (Tokyo, Japan) Glidesheath Slender, in comparison with the currently used 6 French (6 Fr.) radial sheath.

DETAILED DESCRIPTION:
Based on previously reported studies the rates of radial artery occlusion using a standard 6 Fr. sheath is around 5-10%, compared to the single feasibility study of the Glidesheath Slender by Aminian et al (see reference in the citations), the rate of radial artery occlusion was reported 0.88%.

This study will be a prospective randomized, single-blinded (patient-blinded) study, comparing the rate of radial artery occlusion and vascular access site complications between the Glidesheath Slender (Terumo, Tokyo, Japan) and the standard 6 Fr. radial sheath in patients undergoing transradial coronary catheterization.

* The study will enroll patients who will undergo elective or emergency coronary angiography and/or percutaneous coronary intervention (PCI) via transradial approach at the University of Ottawa Heart Institute.
* A baseline clinical vascular & ultrasound assessment will be performed prior to the procedure to document patency of the radial artery.
* Patients will be randomized in 1:1 fashion to either receive the Terumo Glidesheath Slender versus the currently used 6 Fr. sheath.
* The standard angiogram/ PCI will be performed as per usual practice.
* Following the angiogram, clinical vascular assessment as well as an ultrasound will be performed prior to discharge.
* At 30 days follow up the patient will come back for clinical and ultrasound assessment of radial artery patency and access site vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography and/or PCI via transradial approach
* Informed consent
* Documented normal Allen's test

Exclusion Criteria:

* Patient who had a previous angiogram using the same radial artery
* Abnormal Allen's test
* Previous failed radial access.
* Known bleeding disorder or hypercoagulable condition
* Cardiogenic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-03 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | 30 days
  Evaluated clinically and by ultrasound

SECONDARY OUTCOMES:
Vascular access site complications | up to 30 days
  Includes: Radial artery occlusion, bleeding or hematoma, pseudoaneurysm, artery dissection, compartment syndrome of the forearm
Radial artery spasm | participants will be followed for the duration of hospital stay, an expected average of 1 day
Procedure success | participants will be followed for the duration of hospital stay, an expected average of 1 day
  Defined as ability to finish the angiogram/PCI via the intended access site, without the need to change access site.
Sheath kinking | participants will be followed for the duration of hospital stay, an expected average of 1 day
  Major requiring sheath exchange or minor
Painful sheath removal | participants will be followed for the duration of hospital stay, an expected average of 1 day
  Scored on a scale of 1-10 scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Aun-Yeong Chong, MRCP, MD, Principal Investigator — University of Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Kotowycz MA, Johnston KW, Ivanov J, Asif N, Almoghairi AM, Choudhury A, Nagy CD, Sibbald M, Chan W, Seidelin PH, Barolet AW, Overgaard CB, Dzavik V. Predictors of radial artery size in patients undergoing cardiac catheterization: insights from the Good Radial Artery Size Prediction (GRASP) study. Can J Cardiol. 2014 Feb;30(2):211-6. doi: 10.1016/j.cjca.2013.11.021. Epub 2013 Nov 23. PMID 24461923
- [Background] Aminian A, Dolatabadi D, Lefebvre P, Zimmerman R, Brunner P, Michalakis G, Lalmand J. Initial experience with the Glidesheath Slender for transradial coronary angiography and intervention: a feasibility study with prospective radial ultrasound follow-up. Catheter Cardiovasc Interv. 2014 Sep 1;84(3):436-42. doi: 10.1002/ccd.25232. Epub 2013 Nov 6. PMID 24285594
- [Background] Kotowycz MA, Dzavik V. Radial artery patency after transradial catheterization. Circ Cardiovasc Interv. 2012 Feb 1;5(1):127-33. doi: 10.1161/CIRCINTERVENTIONS.111.965871. No abstract available. PMID 22338002